CLINICAL TRIAL: NCT02281162
Title: The Role of Vitamin D and Quetiapine-induced Weight Gain
Brief Title: The Influence of Vitamin D on Atypical Antipsychotic-induced Weight Gain
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: 632260-2
Record Dates: First submitted 2014-09-25; First posted 2014-11-03 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia; Metabolic Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 40 ml venous blood will be collected in three separate tubes. One tube of 10 ml will be sent to the Clinical Pathology Labs for the measurement of complete blood count, complete metabolic panel, fasting lipid profile for the measurement of triglycerides, high density lipoproteins, low density lipoproteins, very low-density lipoproteins. The complete blood count and complete metabolic panel will be done to rule out infection or any other co-morbidity. Another 10 ml tube will be sent to Clinical Pathology lab for the measurement of serum 25-hydroxy D levels. The third tube with 20 ml blood will be used to measure protein and mRNA expression of vitamin D receptor (VDR), CYP24A1 and CYP27B1, and to measure leptin and adiponectin levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weight Gain: No intervention. Will evaluate vitamin D levels and other biomarkers affecting weight with venous blood draw.
  Interventions: Other: Blood Draw
- No Weight Gain: No intervention. Will evaluate vitamin D levels and other biomarkers affecting weight with venous blood draw.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood Draw

SUMMARY:
Schizophrenia and bipolar disorders are major public health problems. The second generation anti-psychotic drugs have efficacy for both positive and negative symptoms and a favorable risk profile as far as movement disorders. However, these drugs are associated with clinically significant weight gain and metabolic effects. The underlying mechanisms of these side effects are unclear, however in our preliminary studies with schizophrenic patients on atypical anti-psychotic drugs, we found that weight gain and vitamin D deficiency was present in about 50% of this population. Given the considerable heterogeneity among the patients on atypical anti-psychotics and potential for weight gain in vitamin D-deficient states, we propose that patients with schizophrenia who gain weight on atypical antipsychotic medications are vitamin D-deficient. This hypothesis will be tested in patients with schizophrenia receiving second-generation anti-psychotic drugs for a minimum duration of 4 months. Specific Aim: We predict that the patients with schizophrenia, who gain weight with antipsychotic treatment, are vitamin D-deficient compared to the patients who do not gain weight. We will examine circulating levels of serum 25(OH)D, mRNA transcripts and protein expression of vitamin D receptor (VDR) and the enzymes, CYP24A and CYP27B, in the white blood cells of the subjects and correlate with BMI and the blood levels of leptin and adiponectin.

DETAILED DESCRIPTION:
Specific Aim: We predict that the patients with schizophrenia, who gain weight with antipsychotic treatment, are vitamin D-deficient compared to the patients who do not gain weight. We will examine circulating levels of serum 25(OH)D, mRNA transcripts and protein expression of vitamin D receptor (VDR) and the enzymes, CYP24A and CYP27B, in the white blood cells of the subjects and correlate with BMI and the blood levels of leptin and adiponectin.

Experimental Approach:

Recruitment of Patients: Subjects will be recruited from the psychiatry clinics of Alegent-Creighton Clinics where the PI is working on a full-time basis. Dr. Selvaraj, the PI of this project, provides psychiatric care annually to an average of 300 patients with schizophrenia and bipolar disorder. In addition, other psychiatrists in the same clinic also see patients with schizophrenia. Thus, there is an ample population available for this study. The patients will be recruited based on the inclusion and exclusion criteria, as shown in Figure 1. Patients with schizophrenia who are on the atypical antipsychotic, quetiapine, will be recruited. The underlying major mechanism of action of this anti-psychotic medication is to block both dopamine (D2 and D4) and serotonin (5-HT2A and 5-HT2c) receptors (24). Also, this antipsychotic medication has been shown to increase weight in the patients. According to the data, mean increase in weight after 8-10 weeks on anti-psychotics is about 12.2 lbs with quetiapine (24). In most cases, increase in weight reaches to a plateau within 8-10 weeks (24). Therefore, we will recruit age-matched patients who have been taking quetiapine 100mg or more for at least 12 weeks. There is no relationship in weight gain and the severity of psychosis or the dose of the anti-psychotic drug. During the first episode, most of these patients are in their 20s and 30s. The patients will be divided into two experimental groups: (i) "Weight gain" and (ii) "No weight gain". In the weight gain group, we will recruit those patients who have gained 10% increase from the baseline weight. In the no weight group, we will recruit patients who have lost weight, did not gain weight or have gained weight <5% over the baseline weight. The baseline weight data and other information will be obtained from the electronic health record through the EPICS system, upon recruitment in the study.

The human research protocol with the Informed Consent and HIPPA forms has been approved by the Institutional Review Board of Creighton University.

Statistical Analysis: The association between weight gain and vitamin D deficiency will be analyzed using 2x2 contingency tables and tests for independence. The three most common tests for independence are the likelihood ratio test (LRT), the Pearson's chi-square statistic, and Fisher's exact test. Both Pearson's chi-square and Fisher's exact test will be used to analyze the data. If the expected number of counts in any one cell is less than five (5), only Fisher's exact test will be reported. The purpose of this pilot is to estimate/confirm a reasonable confidence interval for the true odds ratio and reference proportion to design a larger scale study. We believe we can reasonably recruit between 30 and 40 patients. Should we recruit a total of 40 patients, we believe we can achieve a minimum detectable odds ratio of 9 (with desired power of 0.80 and significance level of 0.05) with reference proportion of 0.35. This initial analysis was based on a preliminary study where 35% of schizophrenic patients gained weight on atypical antipsychotic drugs. Since there is no follow up of these patients, but the collection of the blood and clinical data only at one time point, the question of potential drop-outs or the follow-ups does not arise.

Age-matched subjects of both sex and all ethnicities will participate in this study. Potential subjects will be approached by treating clinicians (inpatient or outpatient) for possible participation; or potential study participants may respond to advertisements in the form of IRB approved flyers that will be distributed at area hospitals and medical clinics. Patients who indicate interest in the study will be asked to sign an informed consent to allow research personnel to review clinical records and speak with the PI or other treating physician about appropriateness for protocol participation. In the Alegent-Creighton clinics we have sufficient number of minority patients, including African-Americans, Hispanics and women. No children will be recruited in this study.

Experimental Protocol: Upon the recruitment of the subjects in this study, the following information will be collected for each of the 40 patients: (i) Demographic data, including age, sex, ethnicity, duration of the illness and the medication regimen and (ii) Anthropometry data, including height, weight, BMI, blood pressure, pulse rate. The following psychiatric rating scale will be used as a diagnostic measure.

The MINI International Neuropsychiatric Interview (M.I.N.I.), a well known psychiatric diagnostic interview protocol, will be administered at baseline before collecting the blood sample. The M.I.N.I. includes items that assess the hallmark symptoms of the exclusionary psychotic depression, other psychotic disorders, bipolar disorder, eating disorder and substance dependence. We will use these modules only to help exclude patients with the prescribed diagnoses.

Following the MINI protocol, 40 ml venous blood, in a fasting state, will be collected in three separate vacutainer EDTA tubes. One tube of 10 ml will be sent to the Clinical Pathology Laboratories for the measurement of complete blood count, complete metabolic panel, fasting lipid profile for the measurement of triglycerides, high density lipoproteins, low density lipoproteins, very low-density lipoproteins. The complete blood count and complete metabolic panel will be done to rule out infection or any other co-morbidity. Another 10 ml tube will be sent to Clinical Pathology lab for the measurement of serum 25-hydroxy D levels. The third tube with 20 ml blood will be used for isolating buffy coat to measure protein and mRNA expression of vitamin D receptor (VDR), CYP24A1 and CYP27B1, and for separating serum to measure leptin and adiponectin levels. This latter part will be done in the research laboratory of the PI using the following procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women with a DSM-IV clinical diagnosis of Schizophrenia, Schizoaffective or Bipolar disorder

  * 21 to 65 years of age; male and female
  * A willingness and ability to provide signed informed consent
  * The subject should have been on quetiapine 100 mg or more for more than 12 weeks.

Exclusion Criteria:

1. Pregnant women
2. Subjects considered at high suicide risk based on the MINI Suicidality Module (> 17 points)
3. Unstable general medical condition or serious illness (e.g. death or hospitalization is anticipated within one year), poor kidney function or liver function (defined as laboratory values ≥ three times the upper limit of the normal), and seizure disorders except for childhood seizure disorders
4. Concurrent therapy with certain psychotropics is permitted, provided that the medication and dose have been stable for the past 90 days
5. Patients on concomitant treatment with clozapine and olanzapine are not permitted.
6. Patients on immunosuppressant medications or any orexigenic or anorexigenic drug
7. Patients on concomitant treatment with amphetamines and/ or methylphenidate
8. History of hypothyroidism or thyroxine therapy
9. Patients with a known condition or undergoing therapeutic measures that affects weight, including but not limited to: eating disorder, type I diabetes, hyperthyroidism, thyroxine therapy, Topamax therapy, and infectious diseases, such as HIV, hepatitis B, and hepatitis C
10. Active supplementation of vitamin D within the last 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: approximately 40 subjects with schizophrenia, bipolar disorder, and schizoaffective disorder, both male and female, 21-65 years, of all ethnicities will be recruited.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Weight Gain in Chart or Graph | less than 12 months
  We expect about 50% patients on anti-psychotic medication will gain weight and these patients will be vitamin D-deficient with <30 ng/ml serum 25(OH)D level.

CONTACTS AND LOCATIONS:
Overall Officials: Vithyalakshmi Selvaraj, MD, Principal Investigator — Creighton University
Locations (1):
- Alegent Creighton Clinic - Psychiatric Associates (Dodge Street), Omaha, Nebraska, United States